CLINICAL TRIAL: NCT02845622
Title: Effects of Hazelnuts and Cocoa on Metabolic Parameters and Vascular Reactivity in Healthy Subjects: A Randomized Controlled Study
Brief Title: Effects of Hazelnuts and Cocoa on Metabolic Parameters and Vascular Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Collaborators: Soremartec Italia S.r.l. (Unknown)
Responsible Party: Principal Investigator, Anna Ferrulli, MD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nocciola/1
Record Dates: First submitted 2016-07-21; First posted 2016-07-27 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Cardiovascular Diseases; Glucose Metabolism Disorders
Keywords: Hazelnut; Cocoa; Flavonoid; Lipids; Vascular Reactivity
MeSH Terms: conditions — Cardiovascular Diseases; Glucose Metabolism Disorders | interventions — Chocolate; Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 30g peeled hazelnuts cream (Experimental): Every person in this group will receive a 30 g peeled hazelnuts cream as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: Hazelnut; Dietary Supplement: Cream
- 30g unpeeled hazelnuts cream (Experimental): Every person in this group will receive a 30 g unpeeled hazelnuts cream as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: Hazelnut; Dietary Supplement: Cream
- snack w/ 30g peeled hazelnuts (Experimental): Every person in this group will receive a snack with 30 g peeled hazelnuts as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: Hazelnut; Dietary Supplement: Snack
- snack w/ 2.5g cocoa powder (Experimental): Every person in this group will receive a snack with 2.5 g cocoa powder as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: Cocoa; Dietary Supplement: Snack
- snack w/ 30g peeled hazelnuts+2.5g cocoa (Experimental): Every person in this group will receive a snack with 30 g peeled hazelnuts and 2.5 g cocoa powder as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: Hazelnut; Dietary Supplement: Cocoa; Dietary Supplement: Snack
- empty snack (Placebo Comparator): Every person in this group will receive an empty snack as an integration to his usual breakfast, and will be asked not to change his diet and physical activity during the 2-week trial.
  Interventions: Dietary Supplement: No hazelnuts / No cocoa; Dietary Supplement: Snack

INTERVENTIONS:
Dietary Supplement: Hazelnut — This dietary supplement contains 30 g of hazelnut.
  Arms: 30g peeled hazelnuts cream; 30g unpeeled hazelnuts cream; snack w/ 30g peeled hazelnuts; snack w/ 30g peeled hazelnuts+2.5g cocoa
Dietary Supplement: Cocoa — This dietary supplement contains 2.5 g of cocoa powder.
  Arms: snack w/ 2.5g cocoa powder; snack w/ 30g peeled hazelnuts+2.5g cocoa
Dietary Supplement: No hazelnuts / No cocoa — This dietary supplement does not contain hazelnut nor cocoa powder.
  Arms: empty snack
Dietary Supplement: Cream — This dietary supplement is just a cream obtained by grinding hazelnuts.
  Arms: 30g peeled hazelnuts cream; 30g unpeeled hazelnuts cream
Dietary Supplement: Snack — This dietary supplement is a commercial snack containing either hazelnut or cocoa or both.
  Arms: empty snack; snack w/ 2.5g cocoa powder; snack w/ 30g peeled hazelnuts; snack w/ 30g peeled hazelnuts+2.5g cocoa

SUMMARY:
This study aims to assess the effects of hazelnuts, cocoa, and the combination of both on vascular reactivity and metabolic profile. Participants, divided in six groups, will receive one of these breakfast integrations for 14 days:

group 1) 30 g peeled hazelnuts;

group 2) 30 g unpeeled hazelnuts;

group 3) snack with 30 g peeled hazelnuts;

group 4) snack with 2.5 g cocoa powder;

group 5) snack with 30 g peeled hazelnuts and 2.5 g cocoa;

group 6) empty snack, control group.

DETAILED DESCRIPTION:
In the last few years, the prevalence of overweight and obesity has increased in all age groups. The European Food Safety Authority stated "cocoa flavanols help maintain endothelium-dependent vasodilation, which contributes to normal blood flow". Several studies reported that a daily consumption of hazelnuts reduces the risk of cardiovascular disease. The hypothesis of this study is to demonstrate a beneficial effect of hazelnut and cocoa diet integrations on vascular reactivity and endocrine-metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-24.9 kg/m2

Exclusion Criteria:

* diabetes mellitus
* glucose intolerance
* dyslipidemia
* metabolic syndrome
* allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effects of a breakfast integration on vascular reactivity, assessed by the variation of peak systolic velocity of the brachial artery, in healthy subjects. | 2 weeks
  Vascular reactivity is measured by assessing the peak systolic velocity (PSV in cm/s) of the brachial artery at rest and after 3 minutes of arterial occlusion using an echographer in Doppler mode. To occlude arterial inflow, a sphygmomanometric cuff is placed above the antecubital fossa and inflated to at least 50 mmHg above systolic pressure for 3 minutes.

SECONDARY OUTCOMES:
Effects of a breakfast integration on total cholesterol (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on high-density lipoprotein-cholesterol (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on low-density lipoprotein-cholesterol (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on triglycerides (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on glucose (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on insulin (uU/mL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on glucagon (pg/mL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on leptin (ng/mL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on ghrelin (ng/mL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on uric acid (mg/dL) in healthy subjects. | 2 weeks
Effects of a breakfast integration on homocysteine (umol/L) in healthy subjects. | 2 weeks
Effects of a breakfast integration on ESR (mm/h) in healthy subjects. | 2 weeks
Effects of a breakfast integration on hs-CRP (mg/dL) in healthy subjects. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- San Donato Hospital, San Donato Milanese, Italy

REFERENCES:
- [Result] Sartori TE, Nunes RA, da Silva GT, da Silva SC, Rondon MU, Negrao CE, Mansur AJ. Influence of demographic and metabolic variables on forearm blood flow and vascular conductance in individuals without overt heart disease. Vasc Health Risk Manag. 2010 Jun 1;6:431-7. doi: 10.2147/vhrm.s10683. PMID 20539845
- [Result] Acree LS, Comp PC, Whitsett TL, Montgomery PS, Nickel KJ, Fjeldstad AS, Fjeldstad C, Gardner AW. The influence of obesity on calf blood flow and vascular reactivity in older adults. Dyn Med. 2007 Mar 26;6:4. doi: 10.1186/1476-5918-6-4. PMID 17386093
- [Result] Papaioannou GI, Seip RL, Grey NJ, Katten D, Taylor A, Inzucchi SE, Young LH, Chyun DA, Davey JA, Wackers FJ, Iskandrian AE, Ratner RE, Robinson EC, Carolan S, Engel S, Heller GV. Brachial artery reactivity in asymptomatic patients with type 2 diabetes mellitus and microalbuminuria (from the Detection of Ischemia in Asymptomatic Diabetics-brachial artery reactivity study). Am J Cardiol. 2004 Aug 1;94(3):294-9. doi: 10.1016/j.amjcard.2004.04.022. PMID 15276091
- [Result] Chandran DS, Jaryal AK, Jyotsna VP, Deepak KK. Impaired endothelium mediated vascular reactivity in endogenous Cushing's syndrome. Endocr J. 2011;58(9):789-99. doi: 10.1507/endocrj.ej11-0030. Epub 2011 Jul 21. PMID 21778615